CLINICAL TRIAL: NCT01937910
Title: Structural and Functional Correlates of Neuroplastic Change Associated With Stroke
Brief Title: Neuroplastic Change in Myelin of the Brain
Acronym: Myelin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H13-01952
Record Dates: First submitted 2013-08-27; First posted 2013-09-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Stroke
Keywords: neuroplastic change; myelin
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stroke Group (Experimental): Participants in the stroke group will complete 10 training sessions of the TRAIT task.
  Interventions: Behavioral: TRAIT Task
- Matched Healthy Control Group (Active Comparator): Participants in the Matched Healthy Control group will complete 10 sessions of the TRAIT task
  Interventions: Behavioral: TRAIT Task

INTERVENTIONS:
Behavioral: TRAIT Task — Increased paretic arm will be manipulated through the performance of a semi-immersive virtual reality-based intercept and release task called TRAIT (TRack And Intercept Task), which is performed in an interactive environment. TRAIT employs an open source Kinect sensor, which tracks 3-D joint movement. Participants are asked to control an on-screen icon using movements of their paretic arm to intercept a moving object as it emerges from the side of a computer screen. Once intercepted, they must accurately throw the object to hit a target. Participants move up through 10 levels of the game as their skill improves. Participants will complete 10 TRAIT training sessions in 4 weeks for a total of 10,000 experimental movements.

SUMMARY:
The main goal of this research is to advance understanding of how stroke changes both the structure and function of the brain. The investigators will determine which is the key driver of recovery of arm function after stroke: changes in the structure of the brain or changes in how brain regions interact with one another.

DETAILED DESCRIPTION:
The main goal of this research is to advance understanding of how stroke changes both the structure and function of the brain. Further, the investigators will determine which is the key driver of recovery of arm function after stroke: changes in the structure of the brain or changes in how brain regions interact with one another. Together, these data will advance the investigators understanding of how neural systems support recovery from stroke. The investigators will use a MRI technique that allows us to assess the health of a brain structure called myelin. This structure is important as it allows information to travel down nerves faster; the more myelin the quicker the signal can be conducted. The investigators aim is to test whether or not movement training can restore myelin in the brain. If movement training does restore myelin in the brain, the investigators will have identified an important new target for rehabilitation interventions.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 40-75
* movement-related deficits associated with a middle cerebral artery stroke
* first time stroke affecting the corona radiata and/or internal capsule
* Fugl-Meyer upper extremity motor score of at least 15 but not greater than 55.

Exclusion Criteria:

* outside the age range of 40-75
* show signs of dementia (score < 24 on the Montreal Cognitive Assessment)
* have aphasia (score < 13 on the Frenchay Aphasia Screen)
* history of head trauma, a major psychiatric diagnosis, neurodegenerative disorder or substance abuse;
* taking any drugs (GABAergic, N-methyl-D-aspartate A-receptor (NMDA) antagonist) known to influence neuroplasticity;
* report contraindications to MRI (see supporting documents)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change in Myelin water fraction | Baseline and 30 days post baseline
  Myelin water fraction (MWF) is the area of the short T2 component (15-35ms) divided by the total T2 distribution expressed as a percentage (MWF% = MWF*100)

SECONDARY OUTCOMES:
Change in Fractional anisotropy | Baseline and 30 days post baseline
  Diffusion properties will be defined by calculating a 6-element tensor ellipsoid to provide both the magnitude and direction of diffusivity in a local orthogonal coordinate system within each voxel. Fractional anisotropy (FA) will be calculated to provide an index of microstructural white matter integrity.

OTHER OUTCOMES:
Change in Hemiparetic arm use measured by accelerometry | Baseline and 30 days post baseline
  Average daily movement counts indexed with accelerometers worn at the wrist

CONTACTS AND LOCATIONS:
Overall Officials: Lara A Boyd, PT; PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided